CLINICAL TRIAL: NCT01992627
Title: A Prospective Randomized Clinical Trial of High Intensity Laser Therapy for Elbow Epicondylosis
Brief Title: Clinical Trial for High Intensity Laser Therapy (HILT) for Elbow Epicondylosis
Acronym: HILT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: CM Chungmu Hospital (Other)
Responsible Party: Principal Investigator, Sang-Hoon Lhee, Director of CM Chungmu Hospital, CM Chungmu Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CMH-2013-01
Record Dates: First submitted 2013-11-12; First posted 2013-11-25 (Estimated); Last update posted 2013-11-25 (Estimated); Status verified 2013-11

CONDITIONS: Chronic Pain; Elbow Tenderness; Elbow Pain Upon Active Resistive Motion
Keywords: High Intensity Laser Therapy; elbow epicondylosis
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- High Intensity Laser Therapy (Experimental): High Intensity Laser Therapy (HILTERAPIA HIRO 3.O)will be used among diagnosed patients with elbow epicondylosis. A five minutes duration of HILTERAPIA HIRO 3.0 along the epicondyle area in a targeted manner will be use on the initial treatment, one week after the initial treatment, two weeks after the initial treatment and four weeks after the initial treatment thereafter.
  Interventions: Device: HILTERAPIA HIRO 3.0

INTERVENTIONS:
Device: HILTERAPIA HIRO 3.0 — High-intensity laser therapy (HILT), which involves higher-intensity laser radiation and which causes minor and slow light absorption by chromophores. This absorption is obtained not with concentrated light but with diffuse light in all directions (the scattering phenomenon), increasing the mitochondrial oxidative reaction and adenosine triphosphate, RNA, or DNA production (photochemistry effects) and resulting in the phenomenon of tissue stimulation called photobiology.

SUMMARY:
This study will determine the efficacy of High Intensity Laser Therapy (HILT) for the treatment of elbow epicondylosis

DETAILED DESCRIPTION:
The diagnosed patients with epicondylosis will be treated with HILTERAPIA HIRO 3.O for a total of four sessions during the entire duration of the treatment protocol. Parameters to be evaluated are tenderness, pain upon active resistive motion and DASH scores. After every treatment session of HILTERAPIA HIRO 3.O, these said parameters will be recorded initially on the first treatment, one week after the initial treatment, two weeks after the initial treatment and four weeks after the initial treatment. Patient is advised to follow-up on the 6th and 12 month post initial HILTERAPIA HIRO 3.O treatment for the reevaluation of the parameters. Tenderness is described as pain upon palpation and is further categorized into, 0= no tenderness, 1 = mild tenderness, 2 = tenderness evident on facial expression and 3 = patient screams upon palpation. Pain is also noted upon active resistive motion of extension/flexion, supination/pronation. Classification includes; 0 = no pain and 1 = mild pain with full power, 2 = severe pain with full power, and 3 = muscle weakness with pain. And for functional scoring will be using the DASH which is a multidimensional disease specific, brief, self-administered measure of symptoms and functional status among subjects with upper limb disorders. The DASH consists of a 30-item questionnaire with 5 response options for each item with a scale ranging from 0, which indicates "least disability," to 100, which indicates "most disability." A change in 12.7 DASH score points is considered to represent clinically significant functional improvement.

ELIGIBILITY:
Inclusion Criteria:

* history of medial and lateral elbow pain for at least three months in duration
* local tenderness for at least three months in duration
* pain on the epicondyle upon active resistive flexion (medial) and extension (lateral) of the wrist

Exclusion Criteria:

* previous elbow conservative managements such as physical therapy and elbow injection-based therapies
* previous surgical management of the elbow

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2013-10; Primary Completion 2013-12 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
DASH as the measure of efficacy for HILT | On the initial treatment, one week after the initial treatment, two weeks after the initial treatment, four weeks after the initial treatment, 6th and 12 month post initial treatment
  The DASH is intended to measure how much difficulty a subject has when performing common functional tasks and activities. The DASH consists of a 30-item questionnaire with 5 response options for each item with a scale ranging from 0, which indicates "least disability," to 100, which indicates "most disability." It incorporates questions related to functional limitations, symptoms, and psychosocial problems. The DASH has been well validated and has a smaller standard error of measurement and a validity comparable to that of joint-specific measures. A change in 12.7 DASH score points is considered to represent clinically significant functional improvement.

SECONDARY OUTCOMES:
Tenderness as the measure of efficacy for HILT | On the initial treatment, one week after the initial treatment, two weeks after the initial treatment, four weeks after the initial treatment, 6th and 12 month post initial treatment
  Tenderness described as pain upon palpation and is further categorized into, 0= no tenderness, 1 = mild tenderness, 2 = tenderness evident on facial expression and 3 = patient screams upon palpation.
Pain upon active resistive motion as the measurement of efficacy for HILT | On the initial treatment, one week after the initial treatment, two weeks after the initial treatment, four weeks after the initial treatment, 6th and 12 month post initial treatment
  Pain is also noted upon active resistive motion of extension/flexion, supination/pronation. Classification includes; 0 = no pain and 1 = mild pain with full power, 2 = severe pain with full power, and 3 = muscle weakness with pain.

CONTACTS AND LOCATIONS:
Overall Officials: Paolo Alan B. Tabar, MD, Principal Investigator — CM Chungmu Hospital
Locations (1):
- CM Chungmu Hospital, Seoul, Yeongdeungpo-gu, South Korea